CLINICAL TRIAL: NCT07363915
Title: A Randomized Controlled Trial Comparing a Manualized Group Program (PADAP) Versus an Active Single-Session Depathologizing Intervention (SSDI) for Subthreshold Anxious-Depressive Symptoms in Primary Care in Spain
Brief Title: Group Program vs Single-Session Depathologizing Intervention for Subthreshold Anxiety-Depression in Primary Care (Spain)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Diego Sanchez Ruiz, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM32-2019-OE18-2019; UAH thesis 1147303 (Other: Universidad de Alcala de Henares); 32/2019 (OE 18/2019) (Other: CEIm Hospital Universitario Príncipe de Asturias)
Record Dates: First submitted 2026-01-02; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Depressive Symptoms; Anxiety Symptoms; Subthreshold Depression
Keywords: Primary Care; Subthreshold Anxiety; Subthreshold Depression; Psychological Intervention; Cognitive Behavioral Therapy; Single-Session Intervention; Randomized Controlled Trial; Depathologizing
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel-group randomized controlled trial comparing PADAP group intervention versus a single-session depathologizing intervention (SSDI).
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment at 12 months was performed by assessors blinded to group assignment. Participants and intervention providers were not blinded. Baseline assessment for the SSDI arm was conducted by the clinician delivering the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PADAP group program (10 sessions) (Active Comparator): Manualized, multimodal, transdiagnostic cognitive-behavioral group intervention delivered in 10 weekly sessions (90 minutes each) by trained clinical psychology residents. Modules cover emotions (psychoeducation), anxiety (physiological arousal management, cognitive restructuring, problem solving), sadness (behavioral activation), and anger (anger regulation and assertiveness training).
  Interventions: Behavioral: PADAP transdiagnostic CBT-based group program
- Single-session depathologizing intervention (SSDI) (Active Comparator): Structured individual single-session intervention (50-60 minutes) delivered by trained clinical psychology residents. The session focuses on empathic listening, shared formulation, contextualization and normalization of distress, narrative reframing (challenging symptoms-as-disease explanations), and activation of personal and social resources outside the healthcare system.
  Interventions: Behavioral: Active Single-Session Depathologizing Intervention (SSDI)

INTERVENTIONS:
Behavioral: PADAP transdiagnostic CBT-based group program — Manualized, multimodal, transdiagnostic cognitive-behavioral group intervention delivered in 10 weekly sessions (90 minutes each) by trained clinical psychology residents. Content includes psychoeducation about emotions; anxiety management (physiological arousal management, cognitive restructuring, problem solving); sadness management (behavioral activation, increasing positive reinforcement); and anger management (anger regulation and assertiveness training).
  Arms: PADAP group program (10 sessions)
Behavioral: Active Single-Session Depathologizing Intervention (SSDI) — Structured individual single-session intervention (50-60 minutes) delivered by trained clinical psychologists/clinical psychology residents. The session focuses on empathic listening and shared formulation; contextualization and normalization of distress; de-pathologizing explanations by challenging symptoms-as-disease narratives; narrative reframing; and activation of personal and social resources outside the healthcare system.
  Arms: Single-session depathologizing intervention (SSDI)

SUMMARY:
This study evaluated two psychological interventions for adults with mild to moderate subthreshold anxious-depressive symptoms in primary care in Spain. Participants referred by general practitioners were randomly assigned to either (1) PADAP, a manualized transdiagnostic group program delivered in 10 weekly 90-minute sessions, or (2) a structured active single-session depathologizing intervention (SSDI), delivered individually in one 50-60-minute session.

The primary aim was to compare changes in depressive and anxiety symptoms from baseline to 12 months. Secondary aims included comparing primary care mental health-related consultations, psychotropic medication use, new contacts with mental health services, and perceived need for further mental health care during follow-up.

DETAILED DESCRIPTION:
This was a prospective, parallel-group randomized controlled trial conducted in four primary care health centres in a large urban area in Spain. Adults aged 18-65 years referred by general practitioners for mild to moderate anxious-depressive symptoms were screened for eligibility. Exclusion criteria included meeting DSM-IV Axis I or II criteria based on the Structured Clinical Interview (SCID-I), current active treatment in mental health services, current substance dependence (except nicotine), organic/neurological/cognitive disorders related to symptoms, or language barriers. All participants provided written informed consent, and the study received ethics approval (reference 32/2019 [OE 18/2019]).

Eligible participants were allocated using a centralized, computerized randomization system to one of two intervention arms. Outcome assessment was performed by a blinded assessor. Participants assigned to SSDI received an individual, structured 50-60-minute session focused on empathic listening, contextualization and normalization of distress, narrative reframing, and activation of personal and social resources outside the healthcare system. Participants assigned to PADAP received a manualized, multimodal, transdiagnostic cognitive-behavioral group intervention delivered in 10 weekly 90-minute sessions covering psychoeducation about emotions and skills to manage anxiety, sadness, and anger.

Depressive symptoms were measured with the Beck Depression Inventory (BDI), and anxiety symptoms with the State-Trait Anxiety Inventory (STAI). Assessments were conducted at baseline and at 12 months. Data on primary care consultations for mental health reasons were extracted from electronic health records, along with information on psychotropic medication use and new contacts with mental health services during follow-up.

ELIGIBILITY:
Inclusion Criteria: 1. Adults aged 18-65 years.

2. Referred from primary care by a general practitioner.

3. Mild to moderate anxious-depressive symptoms based on the GP's clinical judgement during routine consultations, with or without psychotropic medication.

Exclusion Criteria: 1. Meeting DSM-IV Axis I diagnostic criteria based on the Structured Clinical Interview (SCID-I), assessed by two clinical resident psychologists.

2. Receiving active mental health treatment (public or private).

3. Current substance dependence (except nicotine).

4. Organic, neurological, or cognitive disorder related to the symptoms.

5. Language barriers that precluded participation or completion of assessments.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms (STAI-State and STAI-Trait total scores) | Baseline and 12 months
  State-Trait Anxiety Inventory (STAI), State and Trait subscales, total scores. Higher scores indicate greater anxiety symptom severity.
Depressive symptoms (BDI total score) | Baseline and 12 months
  Beck Depression Inventory (BDI), total score. Higher scores indicate greater depressive symptom severity.

SECONDARY OUTCOMES:
GP mental health-related consultations (12 months pre vs 12 months post) | 12 months before intervention and 12 months after intervention
  Number of general practitioner (GP) consultations for mental health reasons extracted from electronic health records (AP Madrid/Horus/HCIS), measured for two periods: (1) the 12 months prior to baseline assessment, and (2) the 12 months following the intervention (post-baseline).
Psychotropic medication use (yes/no) | Baseline and 12 months
  Use of psychotropic medication (antidepressants, anxiolytics, both, or other mood-affecting medication). For analysis, coded as yes/no.
New contact with mental health services (yes/no) | 12 months
  Recorded as yes if the participant requested or received psychological or psychiatric care (public or private) during follow-up.
Perceived need for referral or additional care (yes/no) | 12 months after intervention
  Based on the question: "Do you think you need to be referred to mental health services or receive any other additional intervention from us?". Coded as yes for affirmative responses and for participants who requested referral and were on a waiting list or under follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Sanchez Ruiz, Principal Investigator — University of Alcala
Locations (1):
- Hospital Universitario Príncipe de Asturias (recruitment from 4 primary care centres), Spain, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analysed during the current study are not publicly available due to the risk of compromising participant privacy and because they include information derived from electronic health records, but are available from the corresponding author on reasonable request and subject to approval by the relevant data controller/health service.

REFERENCES:
- See also: Doctoral thesis (protocol and full methods) — http://hdl.handle.net/10017/65579